CLINICAL TRIAL: NCT02974972
Title: Pith Moromo 2: Cohort to Study Health Consequences of Food and Nutrition Insecurity During Pregnancy and Lactation
Acronym: PM2
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Principal Investigator, Sera Young, Assistant Professor, Northwestern University
Other Study IDs: 1405004733
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Food Insecurity; Nutrition; Maternal and Child Health; HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pith Moromo 2 Cohort

SUMMARY:
In this study, the investigators conducted research among HIV-infected and -uninfected pregnant and lactating women to understand the potential role and importance of food insecurity on participant physical and psychosocial health and nutrition.

DETAILED DESCRIPTION:
The central hypothesis of this study was that food and nutrition insecurity are detrimental to the health of HIV+ pregnant women and their infants via nutritional, disease, and psychosocial pathways.

In the first phase, the investigators collected descriptive data to describe and assess food and nutrition insecurity and the associated modifiable determinants among HIV+ pregnant and lactating women in Kenya.

In the second phase, the investigators collected longitudinal cohort data from women who were recruited during pregnancy and have been followed throughout the infant's first year of life.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 years of age with infants
* Infants born to pregnant women enrolled in the cohort study
* HIV-infected pregnant women >18 years of age and ≤30 weeks gestation
* HIV-uninfected pregnant women >18 years of age and ≤30 weeks gestation

Exclusion Criteria:

* Individuals <18 years of age that are not infants born to women enrolled in the cohort study

Ages: 1 Day to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A cohort of 371 pregnant HIV-infected and -uninfected women (ratio 1:1) were recruited from 7 rural and urban clinics in Nyanza, Kenya. Participants were followed from ≤30 weeks pregnancy until 9 months postpartum.
Sampling Method: Non-Probability Sample
Enrollment: 371 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Describing and Assessing the Modifiable Determinants of Food Insecurity (using the Individual Food Insecurity Access Scale) Using A Demography, Health, Nutrition, and Psychosocial Questionnaire at 7 Time Points from Pregnancy to 9 Months Postpartum. | 2 years
  In the first phase the investigators completed descriptive data analysis to describe and assess food and nutrition insecurity and the associated modifiable determinants among HIV+ pregnant and lactating women in Kenya.

SECONDARY OUTCOMES:
Impacts of Food Insecurity (using the Individual Food Insecurity Access Scale) on Maternal and Infant Biomarkers of Health (including anthropometry, hemoglobin, and bioelectrical impedance analysis) | 2 years
  The investigators collected longitudinal cohort data from women who were recruited during pregnancy and have been followed throughout the infant's first year of life. Participants were interviewed at regular intervals and anthropometry and other biomarkers were periodically assessed.
Assessing the Impact of Livestock Ownership on Maternal and Child Health Using Photovoice Qualitative Data Collection Methodology | 1 year
  The investigators collected qualitative data using Photovoice, a participatory photo-elicitation data collection methodology to explore the livestock ownership and perceptions of livestock on household food security (using the Household Food Insecurity Access Scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Evanston, Illinois, United States

REFERENCES:
- [Result] Murnane PM, Miller JD, Tuthill EL, Collins SM, Neilands TB, Onono M, Cohen CR, Weiser SD, Laudenslager ML, Young SL. Perinatal Food Insecurity and Postpartum Psychosocial Stress are Positively Associated Among Kenyan Women of Mixed HIV Status. AIDS Behav. 2020 Jun;24(6):1632-1642. doi: 10.1007/s10461-019-02676-5. PMID 31538283
- [Result] Wang M, Miller JD, Collins SM, Santoso MV, Wekesa P, Okochi H, Onono M, Weiser S, Gandhi M, Young SL. Social Support Mitigates Negative Impact of Food Insecurity on Antiretroviral Adherence Among Postpartum Women in Western Kenya. AIDS Behav. 2020 Oct;24(10):2885-2894. doi: 10.1007/s10461-020-02839-9. PMID 32212069
- [Result] Widen EM, Tsai I, Collins SM, Wekesa P, China J, Krumdieck N, Miller JD, Weiser SD, Onono M, Young SL. HIV infection and increased food insecurity are associated with adverse body composition changes among pregnant and lactating Kenyan women. Eur J Clin Nutr. 2019 Mar;73(3):474-482. doi: 10.1038/s41430-018-0285-9. Epub 2018 Sep 5. PMID 30185898
- [Result] Miller JD, Fitzgerald KG, Smith AL, Young SL. Geophagy among a Cohort of Kenyan Women with Mixed HIV Status: A Longitudinal Analysis. Am J Trop Med Hyg. 2019 Sep;101(3):654-660. doi: 10.4269/ajtmh.19-0149. PMID 31333167
- [Result] Tuthill EL, Miller JD, Collins SM, Widen EM, Onono M, Young SL. HIV infection, hunger, breastfeeding self-efficacy, and depressive symptoms are associated with exclusive breastfeeding to six months among women in western Kenya: a longitudinal observational study. Int Breastfeed J. 2020 Jan 16;15(1):4. doi: 10.1186/s13006-019-0251-8. PMID 31948438
- [Result] Benzaken CL, Miller JD, Onono M, Young SL. Development of a cumulative metric of vaccination adherence behavior and its application among a cohort of 12-month-olds in western Kenya. Vaccine. 2020 Apr 16;38(18):3429-3435. doi: 10.1016/j.vaccine.2020.03.011. Epub 2020 Mar 14. PMID 32184035
- [Derived] Alvarez GG, Miller JD, Santoso MV, Wekesa P, Owuor PM, Onono M, Young SL. Prevalence and Covariates of Food Insecurity Across the First 1000 Days Among Women of Mixed HIV Status in Western Kenya: A Longitudinal Perspective. Food Nutr Bull. 2021 Sep;42(3):319-333. doi: 10.1177/0379572121999024. Epub 2021 May 20. PMID 34011176